CLINICAL TRIAL: NCT06462378
Title: Proton Therapy in Locally Advanced Cervical Cancer in Combination With Concomitant Chemotherapy and Brachytherapy
Brief Title: Proton Therapy for Locally Advanced Cervical Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-22065123
Record Dates: First submitted 2024-05-28; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-05

CONDITIONS: Cervical Cancer; Proton Therapy; Radiotherapy Side Effect
MeSH Terms: conditions — Uterine Cervical Neoplasms; Radiation Injuries | interventions — Proton Therapy

STUDY DESIGN:
Intervention Model Description: Proton therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Proton therapy (Experimental): Proton therapy
  Interventions: Radiation: Proton therapy

INTERVENTIONS:
Radiation: Proton therapy — External beam proton therapy combined with standard cisplatin and brachytherapy

SUMMARY:
The purpose of this protocol is to determine toxicity and efficacy of proton therapy in combination with standard concomitant platinum-based chemotherapy and standard image-guided adaptive brachytherapy (IGABT) in patients with locally advanced cervical cancer (LACC). The over-all aim is to maintain a high disease control and at the same time reduce acute morbidity as well as late side effects after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

  * Cancer of the uterine cervix considered suitable for curative treatment with definitive radio- (chemo) therapy including IGABT
  * Positive biopsy showing squamous-cell carcinoma, adenocarcinoma or adeno-squamous cell carcinoma of the uterine cervix.
  * Staging according to Intenational federation of Gynecology and Obstetrics (FIGO) and TNM guidelines
  * T1-3N1M0 (FIGO stage IIIC1 (with ≥3 pelvic lymph node metastases) and IIIC2)
  * Para-aortic metastatic nodes below L1-L2 are allowed (FIGO stage IVB)
  * Magnetic Resonance Imaging (MRI) and Positron Emission Tomogaraphy-computerized Tomograpy (PET-CT) of the retroperitoneal space and abdomen at diagnosis
  * Patient written, informed consent
  * Age≥18 years
  * Patients must be able to understand a Danish or Swedish

Exclusion Criteria:

* Other primary malignancies except carcinoma in situ of the cervix and basal cell carcinoma of the skin
* Metastatic disease beyond para-aortic region (L1-L2 interspace)
* Previous pelvic or abdominal radiotherapy
* Combination of preoperative radiotherapy with surgery
* Patients receiving neoadjuvant chemotherapy
* Contra indications to MRI
* Contra indications to IGABT
* Contra indications to protontherapy
* Small cell histology (neuroendocrine tumors)
* Active infection or severe medical condition endangering treatment delivery
* Pregnant, lactating or childbearing potential without adequate contraception
* Human Immune Deficiency Virus (HIV)
* Patients with no possibility of follow up

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2029-05-20 (Estimated); Study Completion 2034-05-20 (Estimated)

PRIMARY OUTCOMES:
Acute Bone marrow toxicity | Worst recorded baseline to 3 months after RT
  Grade 2+ Bone marrow toxicity

SECONDARY OUTCOMES:
Late bone marrow toxicity | >3 month to 5 years after RT
  Grade 2+ Bone marrow toxicity
Toxicity | baseline to 5 years after RT
  Toxicity evaluated by NCI-CTCAE v. 5.0 (common terminology criteria for adverse events grade 0-5, 5 indicating worse outcome)
Patient Reported outcomes | baseline to 5 years after treatment
  Patient reported outcomes (by EORTC QLQ-C30, grades 1-4 four indicating worse outcome)
Patient Reported outcomes | baseline to 5 years after treatment
  Patient reported outcomes (by European Organisation for Research and Treatment of Cancer (EORTC) (Quality of life Questionnaire) QLQ-CX24 grades 1-4 four indicating worse outcome)
cisplatin | 3 month
  Cummulative dose (mg)
Oncological outcomes | 5-year
  Progression free survival
Dosimetrics outcomes | 3 month
  External Beam Radiotherapy dose volume to organs at risk (NCI-CTCAE) and comparison to (Image Guided intensity modulated external beam radiochemotherapy and MRI based adaptive brachy therapy in loaclly advanced cervical cancer) EMBRACE II cohort

OTHER OUTCOMES:
Local control | 5-year
  Local tumor control
Overall survial | 5-year
  Overall survial

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Matthiesen, MD, PhD, Principal Investigator — Department of Oncology, Capital Region Denmark
Locations (1):
- Department of Oncology, Capital Region Denmark, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No